CLINICAL TRIAL: NCT03523741
Title: A Clinical Trial to Investigate the Factors Affecting Adverse Drug Reactions and Clinical Efficacy of Clozapine in Korean
Brief Title: Therapeutic Drug Monitoring for Individualized Clozapine Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Euitae Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: CLZ_01
Record Dates: First submitted 2018-05-01; First posted 2018-05-14 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
Keywords: genetic polymorphism; pharmacodynamic variability; personalized pharmacotherapy; adverse drug reaction; quality of life
MeSH Terms: conditions — Schizophrenia; Drug-Related Side Effects and Adverse Reactions | interventions — Clozapine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Clozapine — Clozapine is administered orally according to individual prescribed dosing regimens.
  Other Names: Clozapine treatment

SUMMARY:
The purpose of this study is to evaluate the factors affecting the occurrence of adverse drug reactions (glucose and lipid metabolism abnormality, changes in liver function index and sleeping tendency) and clinical effects in schizophrenia patients with clozapine treatment

DETAILED DESCRIPTION:
1. The baseline tests (sleeping tendency assessment, clinical symptom and cognitive assessments, clinical laboratory tests, genotyping, exploratory biomarker tests, etc.) are conducted to the schizophrenia patients before initiation of the clozapine dosing.
2. On day 15 and 57, the changes from baseline clinical symptom and cognitive function are assessed after clozapine treatment. Also, the occurrence of adverse drug reactions are evaluated. In addition, blood sample collections are performed for the assessment of clozapine and its metabolite levels.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed with schizophrenia spectrum disorder and are expected to use clozapine for more than 57 days to treat or prevent recurrence of schizophrenia
2. Patients who are 19 years or older
3. Patient who understands the contents of the clinical research and provide their written informed consent forms

Exclusion Criteria:

1. Patients taking a drug that the researcher deems inappropriate before clozapine administration
2. Patients who can not use an appropriate contraceptive method during the study period
3. Patients whom the researcher deemed inappropriate for clinical research participation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are diagnosed with schizophrenia spectrum disorder and are expected to use clozapine for more than 57 days to treat or prevent recurrence of schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-13 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Glucose and lipid metabolism abnormality | Change from baseline glucose and lipid profiles on Day 15, and 57
  Change from baseline glucose and lipid profiles after clozapine administration
Liver function abnormality | Change from baseline liver function test on Day 15, and 57
  Change from baseline liver function test
Sleeping tendency assessment | Change from baseline sleeping tendency assessment on Day 15, and 57
  Epworth sleepiness scale (ESS).
  * ESS is comprised of eight questions, each asking about the subject's likelihood of dozing off or falling asleep in a particular situation that is commonly met in daily life.
  * Each ESS item score measures a particular "situational sleep propensity", and respondents use a four-point scale from 0 (no chance of dozing/falling asleep) to 3 (high chance of dozing/falling asleep) for each of the eight questions.
  * The sum of eight item scores (the total ESS score) measures the subject's average sleep propensity across those different situations in daily life. A total ESS score of 16-24 points indicates severe excessive daytime sleepiness.

SECONDARY OUTCOMES:
Cognitive function assessment | Change from baseline MCCB on Day 57, and 127
  MCCB (MATRICS Consensus Cognitive Battery).
Clinical symptom assessment | Change from baseline BPRS on Day 15, and 57
  Brief Psychiatric Rating Scale (BPRS).
  * BPRS is a 24-item scale that measures psychiatric symptoms such as depression, anxiety, hallucinations and unusual behaviour.
  * Each symptom is rated on a scale from 1(not present) to 7(extremely severe).
  * The sum of all 24 items is then calculated to a maximum score of 168. The higher the score, the more psychiatrically impaired the patient is.

OTHER OUTCOMES:
Blood clozapine and its metabolite level | On Day 15, and 57 after clozapine dosing
  Relationship between occurrence of clozapine adverse drug reactions and clozapine blood concentration

CONTACTS AND LOCATIONS:
Overall Officials: Sang-In Park, Ph. D., Study Chair — Kyung Hee University Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided